CLINICAL TRIAL: NCT00501111
Title: A Multi-centre, Double-blind, Double-dummy, Placebo Controlled Parallel Group Randomized Phase IIb Proof of Concept Study With 3 Oral Dose Groups of AZD3480 or Donepezil During 12 Weeks Treatment in Patients With Alzheimer's Disease
Brief Title: Proof of Concept Study of Cognitive Improvement in Patients With Alzheimer's Disease
Acronym: Sirocco
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3690C00010; EuDract 2007-00835-24
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Alzheimer Type; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — ispronicline; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Placebo
- 2 (Active Comparator): donepezil
  Interventions: Drug: Donepezil
- 3 (Experimental): AZD3480
  Interventions: Drug: AZD3480

INTERVENTIONS:
Drug: AZD3480 — 3 oral doses
  Arms: 3
Drug: Donepezil
  Other Names: Aricept
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate that AZD3480 improves cognition in patients with mild or moderate Alzheimer's disease, to assess the safety and tolerability of ZAD3480 and to define the optimal dose(s) to be used in future trials.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent from patient and caregiver
* Clinical prognosis of probable Alzheimer's disease
* Patient must have a caregiver visiting the patient at least three times weekly

Exclusion Criteria:

* Significant neurologic disease or dementia other than Alzheimer's disease
* Major depressive disorder, other major psychiatric disorder
* Use of acetylcholinesterase inhibitor or memantine for treatment of Alzheimer's disease within 8 weeks prior to enrollment
* Impaired vision and/or hearing making cognitive testing difficult

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in ADAS-Cog | assessed after 12 weeks treatment

SECONDARY OUTCOMES:
Change in ADCS-CGIC, Computerized neurological test battery (CDR) and MMSE | assessed after 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AZD3480, Medical Science Director, Study Director — AstraZeneca
Locations (70):
- Austria (4):
  - Research Site, Graz, Osterreich
  - Research Site, Innsbruck, Osterreich
  - Research Site, Vienna, Osterreich
  - Research Site, Linz
- Belgium (5):
  - Research Site, Aalst, Belgium
  - Research Site, Antwerp, Belgium
  - Research Site, Hasselt, Belgium
  - Research Site, Leuven, Belgium
  - Research Site, Sint-Truiden, Belgium
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Ottawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Verdun, Quebec
  - Research Site, Regina, Saskatchewan
- Czechia (10):
  - Research Site, Brno
  - Research Site, Havlíčkův Brod
  - Research Site, Hradec Králové
  - Research Site, Kladno
  - Research Site, Litoměřice
  - Research Site, Nový Jičín
  - Research Site, Olomouc
  - Research Site, Ostrava - Poruba
  - Research Site, Prague
  - Research Site, Prostějov
- Germany (12):
  - Research Site, Bad Saarow
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Freiburg im Breisgau
  - Research Site, Heidelberg
  - Research Site, Kiel-kronshagen
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Nuremberg
- Romania (5):
  - Research Site, Piteşti, Argeş
  - Research Site, Târgu Mureş, Mureș County
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Sibiu
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
- Spain (9):
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Salamanca, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, Hospitalet de Llobregat(barcel, Catalonia
  - Research Site, Salt (girona), Catalonia
  - Research Site, Terrassa, Catalonia
  - Research Site, Madrid, Madrid
  - Research Site, Castellon, Valencia
  - Research Site, Baracaldo (vizcaya)
- United Kingdom (7):
  - Research Site, Uckfield, E Sussex
  - Research Site, Southampton, Hampshire
  - Research Site, Blackpool, Lancashire
  - Research Site, Bradford
  - Research Site, London
  - Research Site, Peterborough
  - Research Site, Swindon

REFERENCES:
- See also: D3690C00010 Clinical Stusy Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=210&filename=D3690C00010.pdf